CLINICAL TRIAL: NCT04179019
Title: Calcium Channel Blockade in Primary Aldosteronism
Acronym: CCB-PA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Anand Vaidya, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P003194
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Primary Aldosteronism; Primary Aldosteronism Due to Adrenal Hyperplasia (Bilateral)
Keywords: primary aldosteronism; calcium channel blocker
MeSH Terms: conditions — Hyperaldosteronism | interventions — Amlodipine

STUDY DESIGN:
Intervention Model Description: Open-label, single group, pilot intervention to evaluate physiologic changes in hormonal parameters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Amlodipine (Experimental): Amlodipine (dose 10 mg, once daily)
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — Amlodipine (10mg daily, as tolerated by blood pressure parameters) for 2 weeks

SUMMARY:
This pilot study explore whether the calcium channel blocker amlodipine can lower aldosterone levels in people with primary aldosteronism.

DETAILED DESCRIPTION:
BACKGROUND:

Primary aldosteronism is a common cause of hypertension. The cause of primary aldosteronism can be a unilateral aldosterone-producing adenoma (APA) or bilateral idiopathic hyperaldosteronism (IHA) whereby there is diffuse production of ectopic and non-physiologic aldosterone in the adrenal cortex. IHA likely contributes to the majority of all primary aldosteronism. Whereas surgical cure is the preferred therapy for APA, lifelong mineralocorticoid receptor antagonists (MRAs), such as spironolactone or eplerenone, are used to treat IHA. Treatment is important as patients with primary aldosteronism have an elevated risk of adverse cardiovascular and renal outcomes compared to patients with essential hypertension. It was long thought that curative surgery and lifelong medical therapy were equivalent treatment options, but more recent studies suggest that MRAs may not ameliorate the adverse cardiovascular and renovascular effects of primary aldosteronism to the same extent as surgery. For one, MRAs do not lower aldosterone levels, in fact, aldosterone levels are often increased with MRA therapy. Therefore, for IHA patients with primary aldosteronism in whom surgery is not an option, efforts to improve and optimize medical therapy are important.

Recent evidence in surgically removed adrenal glands from patients with primary aldosteronism and IHA has shown that even though IHA adrenal glands do not harbor adrenal tumors, they do harbor foci of ectopic aldosterone production and these foci are enriched for somatic mutations (gain of function) in CACNA1D, thereby suggesting that calcium channel mutations are predominant in the pathogenesis of IHA. This represents an intriguing target for medical therapy as blockade of this channel could lower intracellular calcium influx and hence decrease aldosterone production. Calcium channel blockade could also represent a more upstream therapy than mineralocorticoid receptor antagonists, which block the action of aldosterone at its receptor rather than lower its production.

This study is a pilot study to test the hypothesis that calcium channel blockade may lower autonomous aldosterone production in primary aldosteronism patients with IHA.

PROTOCOL:

Participants taking calcium channel blockers will be required to stop these medications for 2-4 weeks prior to initiation of the study. During this time, blood pressure will be managed with doxazosin and/or hydralazine to target an ideal range of <130/80 mmHg, but practically ranges of 120-150/60-90 mmHg will be allowed. Serum potassium will be treated with supplemental potassium chloride to target a range of 3.5-4.5 mEq/L prior to initiation of the study. Participants already on a mineralocorticoid receptor blocker must have a plasma renin activity of <1.0 ng/mL/h to participate, or be able to reduce or stop the dose of this medication for the duration of the study.

Study Visit 1: Participants will be provided sodium supplements (3g/daily) to take for five days prior to study visit 1. On the fifth day, a 24h urine collection will be obtained to measure urinary sodium and aldosterone and participants will arrive at the Clinical Research Center for testing. After one hour of seated rest, baseline blood measures will be obtained, and a single dose of amlodipine 10 mg will be administered. Blood measurements will be repeated every 2 hours to assess the serial change in outcome measures (t=2,4,and 6 hours after the amlodipine dose). Upon completion of the visit, participants will be prescribed amlodipine 10mg daily for 2 weeks.

Treatment phase: Following completion of Visit 1, participants will be prescribed amlodipine 10mg daily for 2 weeks. Home blood pressure monitoring will continue to ensure blood pressure remains in the target range of 120-150/80-90 mmHg. If blood pressure falls below this range with amlodipine, doxazosin and/or hydralazine doses may be reduced or stopped. If blood pressure remains low even after stopping doxazosin and hydralazine, the dose of amlodipine may be lowered to 5mg daily. Potassium chloride supplements may be titrated based on the values obtained at Study visit 1.

Study Visit 2: Participants will be provided sodium supplements (3g/daily) to take for five days prior to study visit 2. On the fifth day, a 24h urine collection will be obtained to measure urinary sodium and aldosterone and participants will arrive at the Clinical Research Center for testing. After one hour of seated rest, baseline blood measures will be obtained, and a single dose of amlodipine 10 mg will be administered. Blood measurements will be repeated every 2 hours to assess the serial change in outcome measures (t=2,4,and 6 hours after the amlodipine dose). Upon completion of the visit, the study will have concluded and participants will return to their usual care.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary aldosteronism
* Idiopathic bilateral hyperaldosteronism subtype based on adrenal venous sampling
* Primary aldosteronism treated with medical therapy (not surgery)
* Plasma renin activity <1.0 ng/mL/h

Exclusion Criteria:

* large or discrete adrenal adenoma on cross-sectional imaging
* inability to stop calcium channel blocker and transition to alternative medication
* inability to stop mineralocorticoid receptor antagonist and transition to alternative medication if plasma renin activity > 1.0 ng/mL/h
* Anemia
* leukopenia
* thrombocytopenia
* pregnant
* breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Vaidya, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Anand Vaidya, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests to share the results of this small pilot study will be considered from clinical researchers with local institutional ethics approval. In these cases, IPD will be shared in a collaborative manner.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after the completion of the study
Access Criteria: clinical researchers with local institutional ethics approval

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the hospital clinics for a diagnosis of known primary aldosteronism
Pre-assignment Details: Prior to assignment, participants taking calcium channel blockers had to to stop these medications for 2-4 weeks. During this time, BP was managed with doxazosin and/or hydralazine to target an ideal range of <130/80 mmHg, but practically ranges of 120-150/60-90 mmHg. In addition, Serum potassium had to be between 3.5-4.5 mEq/L and plasma renin activity had to be <1.0 ng/mL/h, prior to initiation of the study. The inability to achieve these outcomes may result in withdrawal.
Period: Overall Study
Arm/Group | Amlodipine
Started | 15
Completed | 2
Not Completed | 13
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Amlodipine
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 9
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in 24-hour Urinary Aldosterone Excretion Rate
Description: Change in 24h urinary aldosterone excretion rate in response to maximal amlodipine therapy
Time Frame: Baseline and 2 weeks of amlodipine therapy
Measure: Mean (Standard Deviation); unit: mcg/24h
Arm/Group | Amlodipine
Number analyzed (Participants) | 2
mcg/24h | 0.21 (4.94)
Statistical Analysis 1: Comparison: Amlodipine; The intra-individual, paired, 24h urine aldosterone excretion rate following 2 weeks of amlodipine therapy was compared to the baseline pre-treatment 24h urine aldosterone excretion rate. The null hypothesis was that amlodipine therapy would result in no change in the 24h urine aldosterone excretion rate. Because only 2 participants completed the pilot study, the validity of the results is low; Test type: Superiority; p = 0.96, t-test, 2 sided

2. Primary Outcome: Change in Plasma Aldosterone Concentration
Description: Change in plasma aldosterone concentration in response to maximal amlodipine therapy
Time Frame: Baseline and 2 weeks of amlodipine therapy
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Amlodipine
Number analyzed (Participants) | 2
ng/dL | 9.81 (6.87)
Statistical Analysis 1: Comparison: Amlodipine; The intra-individual, paired, plasma aldosterone concentration following 2 weeks of amlodipine therapy was compared to the baseline pre-treatment aldosterone concentration. The null hypothesis was that amlodipine therapy would result in no change in the plasma aldosterone value. Because only 2 participants completed the pilot study, the validity of the results is low; Test type: Superiority; p = 0.29, t-test, 2 sided

3. Secondary Outcome: Acute Change in Plasma Aldosterone Concentration
Description: Change in plasma aldosterone concentration after a single dose of amlodipine, before and after 2 weeks of amlodipine therapy
Time Frame: Baseline plasma aldosterone concentration before amlodipine therapy and 6 hours post-amlodipine dose, compared to baseline plasma aldosterone after 2 weeks of amlodipine therapy and 6 hours post-amlodipine therapy.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Amlodipine
Number analyzed (Participants) | 2
ng/dL | -0.86 (4.51)
Statistical Analysis 1: Comparison: Amlodipine; The intra-individual, paired, change in plasma aldosterone concentration in response to an acute dose of amlodipine (6h post-dose) was compared to the baseline pre-treatment response to an acute dose of amlodipine. The null hypothesis was that an acute amlodipine dose would result in no acute change in the plasma aldosterone levels. Because only 2 participants completed the pilot study, the validity of the results is low; Test type: Superiority; p = 0.83, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: During the course of the study, ranging from 2-8 weeks
Arm/Group | Amlodipine
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine (N=15)
elevated blood pressure (Vascular disorders) | 1 (1)
incidental abnormal labs (Endocrine disorders) | 2 (2) — incidental abnormal labs unrelated to the study procedures or protocol
atypical chest pain unrelated to study protocol (Cardiac disorders) | 1 (1)
hematuria unrelated to the study protocol or procedures (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The major limitations of this pilot study was that it was intended to be a small proof-of-concept study in 15 people with advanced primary aldosteronism given the multi-morbidity nature of this population and difficulty in enrolling them. Further, this was a single-arm study without a control group. Finally, largely influenced by the concurrent COVID pandemic in 2020-2022, only 2 participants completed the pilot study, therefore validity of the results is low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT04179019/Prot_SAP_001.pdf